CLINICAL TRIAL: NCT02480803
Title: Treatment in Advanced Parkinson's Disease: Continuous Intrajejunal Levodopa INfusion VErsus Deep Brain STimulation
Brief Title: INfusion VErsus STimulation in Parkinson's Disease
Acronym: INVEST
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Principal Investigator, J.M. Dijk, J.M. Dijk, MD, PhD, Neurologist, Principal Investigator, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2014_336; 2014-004501-32 (EudraCT Number)
Record Dates: First submitted 2015-05-04; First posted 2015-06-25 (Estimated); Last update posted 2024-02-13 (Actual); Status verified 2024-02

CONDITIONS: Parkinson's Disease
Keywords: Parkinson; Parkinson's Disease; Deep Brain Stimulation; levodopa-carbidopa; Duodopa; continuous intrajejunal infusion
MeSH Terms: conditions — Parkinson Disease | interventions — Deep Brain Stimulation

STUDY DESIGN:
Intervention Model Description: Randomized Clinical Trial
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- continuous levodopa infusion (Active Comparator): continuous intrajejunal infusion of levodopa-carbidopa
  Interventions: Drug: Continuous intrajejunal infusion of levodopa-carbidopa
- deep brain stimulation (Active Comparator): Bilateral deep brain stimulation (DBS) of the subthalamic nucleus (STN)
  Interventions: Device: deep brain stimulation

INTERVENTIONS:
Drug: Continuous intrajejunal infusion of levodopa-carbidopa — Continuous delivery of levodopa-carbidopa intestinal gel through an intrajejunal percutaneous tube (Duodopa, CLI, CILI)
  Other Names: Duodopa infusion; Intestinal levodopa-carbidopa infusion
  Arms: continuous levodopa infusion
Device: deep brain stimulation — Bilateral deep brain stimulation (DBS) of the subthalamic nucleus (STN)
  Other Names: DBS; DBS-STN
  Arms: deep brain stimulation

SUMMARY:
Both Continuous intrajejunal Levodopa Infusion (CLI) and Deep Brain Stimulation (DBS) are accepted therapies for the treatment of advanced Parkinson's disease (PD). To date, no comparative studies have been executed. The INVEST study is an open label randomised controlled trial with cost-effectiveness as primary outcome. The main clinical outcome is quality of life; secondary outcomes are motor symptoms and neurological impairments, among others.

DETAILED DESCRIPTION:
Rationale: Both Continuous intrajejunal Levodopa Infusion (CLI) and Deep Brain Stimulation (DBS) are accepted therapies for the treatment of advanced Parkinson's disease (PD). As directly comparative studies are lacking, it is unknown whether one of the therapies is more effective. Besides, CLI seems to be more expensive. To determine the optimal treatment in advanced PD, a comparative study of CLI and DBS is warranted.

Hypothesis: We hypothesize that CLI is a more expensive therapy in advanced PD than DBS and that the surplus in costs is not cost-effective with regard to benefits for the patient and caregivers in quality of life, PD symptoms and adverse events.

Objective: To realize a cost-effective treatment strategy in advanced PD. Study design: Prospective, randomized, open label multicentre trial, with two additional patient preference treatment arms ("patient preference randomized trial").

Study population: Patients with PD who, despite optimal pharmacological treatment, have severe response fluctuations, dyskinesias, painful dystonia, or bradykinesia. A total of 66 patients will be randomized, at least 120 patients will be included in the patient preference arms.

Intervention: Patients will be randomized to DBS or CLI. For DBS treatment, 2 electrodes will be implanted in the brain. The electrodes are connected to an implanted pulse generator, which will be placed subcutaneously in the subclavian area. For CLI treatment, a tube will be placed in the jejunum via a percutaneous endoscopic gastrostomy (PEG). This tube is connected to an external pump that delivers the levodopa-gel.

Main study parameters: There are 8 specified assessment visits: at baseline, and 1 week, 3, 6, 9, 12, 24 and 36 months after start of the study treatment. The primary health economic outcomes are the costs per changed unit on the PDQ-39 (and the costs per changed QALY for the cost-effectiveness and cost-utility analyses, respectively. The EQ-5D will be applied as the utility measure. Change in quality of life (expressed in the between group difference in change from baseline to 12 months on the PDQ-39 summary index score) is the main clinical outcome. Among the secondary outcomes are functional health, complications and adverse effects, use of care and perceptions of patients and neurologists regarding both treatments.

ELIGIBILITY:
Inclusion Criteria:

* Idiopathic Parkinson's Disease with bradykinesia and at least two of the following signs; resting tremor, rigidity, and asymmetry;
* Despite optimal pharmacological treatment, at least one of the following symptoms: severe response fluctuations, dyskinesias, painful dystonia or bradykinesia;
* A life expectancy of at least two years.

Exclusion Criteria:

* Age below 18 years
* Previous PD-neurosurgery (e.g., DBS, pallidotomy, thalamotomy);
* Previous CLI (through a PEG-tube or Nasal Jejuna| tube);
* Hoehn and Yahr stage 5 at the best moment during the day;
* Other severely disabling disease;
* Dementia or signs of severe cognitive impairment
* Psychosis;
* Current depression;
* Contraindications for DBS surgery, such as a physical disorder making surgery hazardous;
* Contraindications for PEG surgery such as interposed organs, ascites and oesophagogastric varices, or for Duodopa;
* Pregnancy, breastfeeding, and women of child bearing age not using a reliable method of contraception;
* No informed consent;
* Legally incompetent adults;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2014-12-19 (Actual); Primary Completion 2021-12-07 (Actual); Study Completion 2024-01-26 (Actual)

PRIMARY OUTCOMES:
Cost effectiveness in costs per changed unit on PDQ-39 | 12 months
  The costs per changed unit on the PDQ-39.
Cost-utility in costs per changed Quality Adjusted Life Year (QALY, years) | 12 months
  The costs per QALY. The EuroQol 5D-3L (EQ-5D; 5 questions, each score 1-3, providing a health state, to be translated with provided Valuation set) will be applied as the utility measure.

SECONDARY OUTCOMES:
Quality of life (on PDQ-39) | 12, 24 and 36 months
  Changes from Baseline on Parkinson's Disease Questionnaire-39 (PDQ-39; score 0-100, higher score is lower quality of life)
Quality of life (on EQ-5D) | 12, 24 and 36 months
  Change from Baseline on EuroQol 5D-3L (EQ-5D; 5 questions, each score 1-3, providing a health state, to be translated with provided Valuation set)
Motor symptoms | 12 and 36 months
  Score changes from Baseline in off and on state on Movement Disorder Society's Unified Parkinson Disease Rating Scale (MDS-UPDRS part 3; 0-132, high score is more motor symptoms)
Motor symptoms: time in off and on-state | 12, 24 and 36 months
  Change from Baseline in time in off-state, on-state without dyskinesias, on-state without troublesome dyskinesias and on-state with troublesome dyskinesias measured with motor symptom diary
Motor experiences of daily living | 12, 24 and 36 months
  Changes from Baseline on MDS-UPDRS part 2 (Movement Disorder Society's Unified Parkinson Disease Rating Scale (MDS-UPDRS part 2; score 0-52, high score is more worse health)
Dyskinesia | 12 and 36 months
  Change from Baseline on clinical Dyskinesia Rating Scale (CDRS; score 0-28, high score is more dyskinesia)
PD-medication (levodopa-equivalent dose) | 12, 24 and 36 months
  Change from Baseline expressed in levodopa-equivalent dose
Functional health status | 12, 24 and 36 months
  Change from Baseline on Amsterdam Linear Disability Score (ALDS, 29 items; 0-100, high score is high level of functional status)
Non-motor symptoms (Non Motor Symptom Checklist) | 12, 24 and 36 months
  Changes from Baseline on Non Motor Symptom Checklist
Non-motor symptoms (Rotterdam Symptom Checklist | 12, 24 and 36 months
  Change from Baseline on Rotterdam Symptom Checklist
Non-motor symptoms (SCOPA-AUT) | 12, 24 and 36 months
  Change from Baseline on SCOPA-AUT (SCales for Outcomes in PArkinson's Autonomic symptoms; score 0-92, higher score is more symptoms)
Disability | 12, 24 and 36 months
  Change from Baseline in Hoehn and Yahr stage (H&Y stage; 1-5: a higher score is more disease progression)
Cognitive functioning | 12 and 36 months
  Change from Baseline on Parkinson's Disease Cognition Rating Scale (PD-CRS; 0-134, higher score is a result of better cognitive performance)
Cognitive functioning Mattis | 12 and 36 months
  Change from Baseline in Mattis Dementia Rating score (score 0-144, higher score is better cognitive function)
Neuropsychologic functioning BNT | 12 and 36 months
  Change from Baseline in Boston Naming Test (range 0-30, higher is better)
Neuropsychologic functioning Letter Fluency | 12 and 36 months
  Change from Baseline in Letter Fluency (score 0-100, higher is better)
Neuropsychologic functioning WAIS IV | 12 and 36 months
  Change from Baseline in WAIS IV (Wechsler Adult Intelligence Scale IV - subsection similarities; score 0-36, higher is better)
Neuropsychologic functioning Reading | 12 and 36 months
  Change from Baseline in Dutch Reading Test (0-100, higher is better)
Neuropsychologic functioning Word Test | 12 and 36 months
  Change from Baseline in 15 word test (0-75, higher is better)
Neuropsychologic functioning Memory | 12 and 36 months
  Change from Baseline in Rivermead Behavioral memory test (subsection stores; score 0-42, higher is better)
Neuropsychologic functioning Trail making | 12 and 36 months
  Change from Baseline in Trail making test (score 10-500, higher score is longer time, i.e. worse score)
Neuropsychologic functioning Color Word | 12 and 36 months
  Change from Baseline in Stroop Color Word Test (score 10-1000, higher is better)
Neuropsychologic functioning Line Orientation | 12 and 36 months
  Change from Baseline in Judgement of line orientation (score 0-30, higher is better)
Neuropsychologic functioning Clock | 12 and 36 months
  Change from Baseline in Clock construction (score 0-14, higher is better)
Psychiatric disease | 12 and 36 months
  Change from Baseline in Mini International Neuropsychiatric Interview
Apathy | 12, 24 and 36 months
  Change from Baseline in Starkstein's Apathy Scale (SAS; score 0-42, high score is more signs of apathy)
Compulsive Disorders | 12, 24 and 36 months
  Change in presence of Compulsive Disorder from Baseline assessed with Parkinson's Disease Impulsive-Compulsive Disorders Questionnaire (QUIP, utilizing established thresholds)
Anxiety | 12 and 36 months
  Changes from Baseline on Hamilton Anxiety Scale (HAM-A; 0-56, high score is worse outcome)
Depression | 12 and 36 months
  Change from Baseline on Hamilton Depression Rating Scale (HDRS; 0-68, higher score is worse outcome)
Suicidality | 12 and 36 months
  Changes from Baseline on Columbia Suicide Severity Rating Scale (range 0-25, higher score is worse outcome)
Adverse effects | 12, 24 and 36 months
  Number of participants with adverse effects and description of these
Complications and description of complications | 12, 24 and 36 months
  Number of participants with complications and description of these
Stopping allocated treatment | 12, 24 and 36 months
  Number of participants who stopped treatment
Treatment failure | 12, 24 and 36 months
  Number of participants with treatment failure
Treatment cross-over | 12, 24 and 36 months
  Number of participants with treatment cross-over
Patient satisfaction | 12, 24 and 36 months
  Descriptive questionnaire, no scale applied, descriptive statistics
Patients attitude to treatment | 12, 24 and 36 months
  Change from Baseline on Patient Reported Outcome Scale (range 0-128, high score is worse outcome)
Medical costs | 12, 24 and 36 months
  Calculation of the total costs in euro by means of iMCQ (iMTA Medical Consumption Questionnaire)
Non-medical care costs | 12, 24 and 36 months
  Calculation of the total costs in euro by means of iPCQ (iMTA Productivity Cost Questionnaire)
Caregiver burden | 12, 24 and 36 months
  Descriptive questionnaire, no scale applied, descriptive statistics

CONTACTS AND LOCATIONS:
Overall Officials: Joke M Dijk, MD, PhD, Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Locations (1):
- Academic Medical Center, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] van Poppelen D, Sisodia V, de Haan RJ, Dijkgraaf MGW, Schuurman PR, Geurtsen GJ, Berk AEM, de Bie RMA, Dijk JM. Protocol of a randomized open label multicentre trial comparing continuous intrajejunal levodopa infusion with deep brain stimulation in Parkinson's disease - the INfusion VErsus STimulation (INVEST) study. BMC Neurol. 2020 Jan 31;20(1):40. doi: 10.1186/s12883-020-1621-y. PMID 32005175

DOCUMENTS (2):
  • Study Protocol (2019-10-07): https://cdn.clinicaltrials.gov/large-docs/03/NCT02480803/Prot_000.pdf
  • Statistical Analysis Plan (2022-03-18): https://cdn.clinicaltrials.gov/large-docs/03/NCT02480803/SAP_001.pdf